CLINICAL TRIAL: NCT00006257
Title: Phase I Trial of SU5416 in Combination With Weekly Paclitaxel in Patients With Advanced Malignancies
Brief Title: SU5416 and Paclitaxel in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068191; U01CA062505 (NIH); P30CA033572 (NIH); CHNMC-PHI-30; CHNMC-IRB-99098; NCI-T99-0086
Record Dates: First submitted 2000-09-11; First posted 2003-10-08 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Paclitaxel; Semaxinib

INTERVENTIONS:
Drug: paclitaxel
Drug: semaxanib

SUMMARY:
RATIONALE: Drugs such as SU5416 may stop the growth of cancer by stopping blood flow to the tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining SU5416 with chemotherapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining SU5416 and paclitaxel in treating patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of SU5416 when combined with paclitaxel in patients with advanced malignancies.
* Determine the toxicities and pharmacokinetics of this regimen in these patients.
* Determine the effects of this regimen on a variety of histological and molecular biomarkers of angiogenesis, including in vitro activity assays of endothelial cell proliferation, migration, and invasion.

OUTLINE: This is a dose escalation study of SU5416.

Patients receive SU5416 IV over 1 hour twice weekly during the first week. During subsequent courses, SU5416 is administered on days 1, 4, 8, 11, 15, 18, 22, and 25. Paclitaxel begins on the second week of therapy and is administered IV over 1 hour on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of SU5416 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: Approximately 24 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven advanced malignancy for which no satisfactory treatment exists
* Must have tumor accessible by biopsy

  * Minimum of 1 baseline biopsy required
* No brain metastases or primary CNS tumor

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* SGOT and SGPT less than 2 times upper limit of normal unless due to presence of tumor
* Bilirubin normal

Renal:

* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No uncompensated coronary artery disease by ECG or physical examination
* No myocardial infarction or severe unstable/angina within the past 6 months
* No severe peripheral vascular disease associated with diabetes mellitus
* No severe deep vein or arterial thrombosis within the past 3 months

Pulmonary:

* No pulmonary embolism within the past 3 months

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No unstable or severe concurrent medical condition
* No active uncontrolled infection
* No history of allergic reaction to paclitaxel or Cremophor
* No greater than grade 1 peripheral neuropathy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior SU5416

Chemotherapy:

* No prior paclitaxel
* Greater than 4 weeks since prior chemotherapy (6 weeks for nitrosourea or mitomycin) and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* Greater than 4 weeks since prior radiotherapy and recovered

Surgery:

* See Disease Characteristics

Other:

* Recovered from any prior investigational agents
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-11

CONTACTS AND LOCATIONS:
Overall Officials: Przemyslaw W. Twardowski, MD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California